CLINICAL TRIAL: NCT02934529
Title: A Randomised Study to Assess the Efficacy of Cetuximab Rechallenge in Patients With Metastatic Colorectal Cancer (RAS Wild-type) Responding to First-line Treatment With FOLFIRI Plus Cetuximab
Brief Title: Metastatic Colorectal Cancer (RAS-wildtype) After Response to First-line Treatment With FOLFIR Plus Cetuximab
Acronym: AIO-KRK-0114
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, PD Dr. med. Volker Heinemann, Director of the Comprehensive Cancer Center (CCCLMU), Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIRE-4; 2014-003787-21 (EudraCT Number)
Record Dates: First submitted 2015-03-19; First posted 2016-10-17 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Leucovorin; Fluorouracil; Cetuximab; Bevacizumab; Capecitabine; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- A1 (Active Comparator): FOLFIRI plus cetuximab: one cycle (cycle duration 14 days) consists of Irinotecan, Folinic acid 5-FU, cetuximab
  Administration every two weeks until progression in first-line or emergence of unacceptable toxicity.
  De-escalation (e.g. to irinotecan plus cetuximab or FUFA plus cetuximab) is allowed, but cetuximab should be administered until progression if safety is adequate.
  Interventions: Drug: Irinotecan; Drug: Folinic Acid; Drug: 5-FU; Drug: Cetuximab
- B1 (Experimental): FOLFIRI plus cetuximab: one cycle (cycle duration 14 days) consists of Irinotecan, Folinic acid 5-FU, cetuximab
  Administration every 2 weeks for a maximum of 12 cycles
  * Treatment may be de-escalated to irinotecan plus cetuximab or FUFA plus cetuximab, prior to 12 cycles, for toxicity if necessary, if the best response has been SD,
  * Treatment may undergo 'switchover' to a fluoropyrimidine and bevacizumab, between 8 and 12 cycles, for toxicity if necessary, if the best response has been CR or PR,
  Interventions: Drug: Irinotecan; Drug: Folinic Acid; Drug: 5-FU; Drug: Cetuximab
- B1 Switchover regimens (Experimental): Switchover to FUFA plus bevacizumab every three weeks (cycle duration 21 days) until progression in first-line or emergence of unacceptable toxicity.
  Folinic acid, 5-FU, Bevacizumab
  1st administration 90 min. in case of good safety, the second 60 min. further administration 30 min.
  Or alternatively Switchover to capecitabine plus bevacizumab every three weeks (cycle duration 21 days) until progression in the first-line or emergence of unacceptable toxicity.
  Interventions: Drug: Folinic Acid; Drug: 5-FU; Drug: Bevacizumab; Drug: Capecitabine
- A2 (third line) (Active Comparator): Treatment at the treating physician's discretion depending on the patient's general condition, with the exclusion of any anti-EGFR treatment whatsoever (such as for example cetuximab, panitumumab). Recommendations include Regorafenib in line with Grothey A et al, Lancet. 2013
  or alternatively another anti-EGFR-free treatment according to the investigating physician's choice
  Administration until progression occurs in the third line or unacceptable toxicity
  Interventions: Drug: regorafenib
- B2 (third line) (Experimental): one cycle (cycle duration 14 days) consists of Irinotecan 125mg, Folinic acid, 5-FU, cetuximab wkly
  Administration every 2 weeks until progression occurs in the third line or unacceptable toxicity
  or depending on the patient's general condition and the study physician's decision
  Irinotecan plus cetuximab in line with Cunningham D et al, N Engl J Med. 2004
  Interventions: Drug: Irinotecan; Drug: Folinic Acid; Drug: 5-FU; Drug: Cetuximab; Drug: Irinotecan 125mg; Drug: Cetuximab wkly

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 180 mg/m² iv, 30 - 90 min., day 1, q d15
  Other Names: Campto
  Arms: A1; B1; B2 (third line)
Drug: Folinic Acid — Folinic acid (racemic) 400 mg/m² iv, 120 min. day 1, q d15
  Other Names: Folgamma mono
  Arms: A1; B1; B1 Switchover regimens; B2 (third line)
Drug: 5-FU — 5-FU 400 mg/m² bolus day 1, q d15
  Other Names: Fluorouracil
  Arms: A1; B1; B1 Switchover regimens; B2 (third line)
Drug: 5-FU — 5-FU 2400 mg/m² iv over 46 h day 1-2, q d15
  Other Names: Fluorouracil
  Arms: A1; B1; B1 Switchover regimens; B2 (third line)
Drug: Cetuximab — cetuximab initially 400 mg/m² as a 120 min. infusion (≤ 5mg/min); subsequently 250 mg/m² iv respectively as a 60 min. infusion (≤ 10mg/min) day 1 + 8
  Other Names: Erbitux
  Arms: A1; B1; B2 (third line)
Drug: Bevacizumab — Bevacizumab 7.5 mg/kg BW iv over 30 to 90 minutes: day 1
  Other Names: Avastin
  Arms: B1 Switchover regimens
Drug: Capecitabine — Capecitabine 1250 mg/m2 2 x day p.o. day 1-14, q d15
  Other Names: Xeloda
  Arms: B1 Switchover regimens
Drug: regorafenib — 160 mg per day (day 1-21) (repeated on day 28)
  Other Names: CAS #:755037-03-7
  Arms: A2 (third line)
Drug: Irinotecan 125mg — Irinotecan 125 mg/m² iv, 60 - 90 min. weekly (D1, D8, D15, D22)
  Other Names: Campto
  Arms: B2 (third line)
Drug: Cetuximab wkly — Cetuximab initially 400 mg/m² as a 120 min. infusion (≤ 5mg/min); subsequently 250 mg/m² iv respectively as a 60 min. infusion (≤ 10mg/min) weekly (D1, D8, D15, D22, D29, D36)
  Other Names: Erbitux
  Arms: B2 (third line)

SUMMARY:
The FIRE-4 study aims to define a treatment concept for patients with RAS wild-type tumours, optimised with regard to overall survival. The first-line treatment will be conducted with FOLFIRI plus cetuximab, which resulted in a significantly prolonged overall survival versus bevacizumab in the FIRE-3 study. Following initial progression (PD1) it is recommended that the treatment be continued with FOLFOX plus bevacizumab, as this concept led to significantly prolonged survival in the E3200 study. Owing to the encouraging results of the Santini study , a cetuximab rechallenge in combination with irinotecan-based chemotherapy is to be performed as part of the third-line treatment in patients who showed a response defined according to RECIST 1.1 during the first-line treatment (tumour diameter < -30%) or presented with stable tumour disease for at least 6 months (tumour diameter +20 to -30%). The concept of the ideal sequence has not yet been studied to date in a clinical trial.

DETAILED DESCRIPTION:
The study will begin with FPFV: (first study visit of the first patient, signing the declaration of consent to participate in the study): scheduled for the 4th quarter of 2014

Patient recruitment: 36 months

Treatment duration per patient: Until the time of progression under the third-line treatment at the latest. Anticipated individual duration of treatment: 24 months (for patients who undergo all three treatment lines -included in part 1), or 6 months in patients who only receive third line treatment (included directly in part 2)

Duration of follow-up after the end of treatment: For all patients, until death or for at least 1 year following final termination of any study treatment regardless of the treatment line. In so doing, the follow-up period for patients included in part 1 of the study will be conducted for a maximum of 5 years from the time of randomisation 1; and for patients included in only part 2 of the study (third-line treatment), for a maximum of 3 years from the date of randomisation 2.

End of the study: last follow-up visit of the last study patient scheduled for the 4th quarter of 2020

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, UICC stage IV adenocarcinoma of the colon or rectum (metastatic colorectal cancer), primarily nonresectable or with surgery refused by the patient
* RAS wild-type tumour status (KRAS and NRAS exon 2-4) (proven in the primary tumour or metastasis) at any timepoint of randomisation
* Age ≥18
* ECOG performance status 0-1
* Patients suitable for chemotherapy administration
* Patient's written declaration of consent obtained
* Estimated life expectancy > 3 months
* Presence of at least one measurable reference lesion according to the RECIST 1.1 criteria (chest and abdominal CT 4 weeks or less before randomisation)
* Primary tumour tissue available and patient consents to storage and molecular and genetic profiling of blood, plasma and tumour material (patients included directly at Part 2 of the study in whom primary tumour material is no longer available may be included in the study, provided that tumour material from the compulsory biopsy on progression following second-line treatment is available).
* Effective contraceptive measures in men and in women of childbearing age (Pearl index <1)
* Adequate haematopoietic function:

  * Leukocytes ≥ 3.0 x 109/L with neutrophils ≥ 1.5 x 109/L
  * Thrombocytes ≥ 100 x 109/L,
  * Haemoglobin ≥ 5.6 mmol/L (equivalent to 9 g/dL)
* Adequate hepatic function:

  * Serum bilirubin ≤ 1.5 x upper normal limit,
  * ALAT and ASAT ≤ 2.5 x upper normal limit (in the presence of hepatic metastases, ALAT and ASAT ≤ 5 x upper normal limit)
* INR < 1.5 and aPTT < 1.5 x upper normal limit (patients without anticoagulation). Therapeutic anticoagulation is allowed if INR and aPTT have remained stable within the therapeutic range for at least 2 weeks.
* Adequate renal function:

  * Serum creatinine ≤ 1.5 x upper normal limit or creatinine clearance (calculated according to Cockcroft and Gault) ≥ 50ml/min.
* adequate cardiac function: ECG and echocardiogram with a LVEF of ≥55%
* Any significant toxicities of previous treatments must have resolved or stabilised
* Last administration of an anti-EGFR substance ≥ 4 months before randomisation 2

Inclusion criterion solely for Part 1:

* No previous chemotherapy for metastatic disease
* Time since last administration of a previous adjuvant chemotherapy >6 months

Additional inclusion criteria solely for Part 2:

* Former first-line treatment of the metastatic colorectal cancer with FOLFIRI and cetuximab; data available for the duration of treatment and the response within the context of first-line treatment
* Former second-line treatment of the colorectal cancer without FOLFIRI, irinotecan or an anti-EGFR substance with data available for the substances administered, duration of treatment and response within the context of the second-line treatment
* Proof of a RAS wild-type tumour (KRAS and NRAS exons 2-4) in a tumour biopsy (metastasis) within 4 weeks before randomisation
* CT examinations with evidence of a partial response (PR) or complete response (CR) or stable disease (SD) ≥6 months according to RECIST Version 1.1 criteria as best response within the context of the first-line treatment with FOLFIRI and cetuximab

Exclusion Criteria:

* Proof of a RAS mutation (KRAS or NRAS, exons 2-4 in the tumour (proven in the primary tumour or metastasis) or absence of testing for RAS mutation
* Primarily resectable metastases and the patient wishes for resection
* Grade III or IV heart failure (NYHA classification)
* Myocardial infarction, unstable angina pectoris, balloon angioplasty (PTCA) with or without stenting within the past 12 months before inclusion in the study
* Pregnancy (exclusion to be ascertained by a beta hCG test) or breast feeding
* Medical or psychological impairments associated with restricted ability to give consent or not allowing conduct of the study
* Additional cancer treatment (chemotherapy, radiation, immune therapy or hormone treatment) during the study treatment in first-line and third-line treatment (treatments that are conducted as part of an anthroposophic or homeopathic treatment approach, e.g. mistletoe therapy do not represent an exclusion criterion)
* Previous chemotherapy for the colorectal cancer with the exception of adjuvant treatment, completed at least 6 months before entering the study (exclusion criterion solely for part 1)
* Participation in a clinical study or experimental drug treatment within 30 days prior to inclusion or during participation in the study
* Known hypersensitivity or allergic reaction to any of the following substances: 5-fluorouracil, cetuximab, oxaliplatin, irinotecan, bevacizumab and chemically related substances
* Known or clinically suspected brain metastases
* History of acute or subacute intestinal occlusion or chronic inflammatory bowel disease or chronic diarrhoea
* Symptomatic peritoneal carcinosis
* Severe, non-healing wounds, ulcers or bone fractures
* Uncontrolled hypertension
* Marked proteinuria (nephrotic syndrome)
* Arterial thromboemboli or severe haemorrhage within 6 months prior to inclusion in the study (with the exception of tumour bleeding before tumour resection surgery)
* Haemorrhagic diathesis or tendency towards thrombosis
* Known DPD deficiency (specific screening not required)
* Known glucuronidation deficiency (Gilbert's syndrome) (specific screening not required)
* History of a second malignancy during the past 5 years before inclusion in the study or during participation in the study, with the exception of a dermal basal cell or squamous cell carcinoma or cervical carcinoma in situ, if these were treated curatively.
* Known history of alcohol or drug abuse
* A significant concomitant disease which, in the investigating physician's opinion, rules out the patient's participation in the study
* Absent or restricted legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2015-03; Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival | up to 55 months
  overall survival from randomisation to third-line treatment (OS3) under cetuximab rechallenge versus an anti-EGFR-free treatment in patients responding to treatment with cetuximab

SECONDARY OUTCOMES:
Response Rate | up to 55 months
  Response rate ORR1, 2 & 3 (assessment of ORR 1 and ORR 2 only if the patient was already included in part 1 of the study)
Progression-free survival | up to 55 months
  Progression-free survival PFS1, 2 & 3 (assessment of PFS 1 and PFS 2 only if the patient was already included in part
  1 of the study)
Overall Survival (first-line treatment) | up to 55 months
  Overall survival (OS1) from randomisation to first-line treatment (assessment only if the patient was already included in part 1 of the study)
Depth of Response | up to 55 months
  Investigation of depth of response during first-line treatment and third-line treatment.
Early tumor shrinkage | up to 55 months
  Investigation of early tumour shrinkage during first-line treatment and third-line treatment.
molecular biomarkers | up to 67 months
  Study of molecular biomarkers for prediction of sensitivity and secondary resistance to an anti-EGFR treatment with cetuximab (including tumour biopsies and liquid biopsies from blood samples)
Biomarker Score | up to 67 months
  Prospective validation of a biomarker score (RAS and BRAF)
tumour marker | up to 55 months
  Prospective analysis of tumour marker evolution (CEA and CA 19-9)
Safety and tolerance as measured by the NCI-CTCAE version 4.03 criteria | up to 55 months
  Recording of the safety and tolerance (NCI-CTCAE version 4.03 criteria) of the first-line and third-line treatment

CONTACTS AND LOCATIONS:
Overall Officials: Volker Heinemann, Prof. Dr., Principal Investigator — Maximilians University of Munich, Comprehensive Cancer Center and Medical Dept. III
Locations (1):
- Klinikum der Universitaet Muenchen - Campus Grosshadern, Munich, Germany

REFERENCES:
- [Derived] Stintzing S, Klein-Scory S, Fischer von Weikersthal L, Fuchs M, Kaiser F, Heinrich K, Modest DP, Hofheinz RD, Decker T, Gerger A, Angermeier S, Rumpold H, Dickhut A, Ohler L, Gruenberger B, Niedersuess-Beke D, Sandmann M, Winder T, Trojan J, Prager G, Held S, Kumbrink J, Schmiegel W, Baraniskin A, Heinemann V. Baseline Liquid Biopsy in Relation to Tissue-Based Parameters in Metastatic Colorectal Cancer: Results From the Randomized FIRE-4 (AIO-KRK-0114) Study. J Clin Oncol. 2025 Apr 20;43(12):1463-1473. doi: 10.1200/JCO.24.01174. Epub 2025 Feb 4. PMID 39903881